CLINICAL TRIAL: NCT02716961
Title: Prospective Cohort Study of Transurethral Resection of Bladder Tumor (TURBT) Combined With Adjuvant Intravenous GC Chemotherapy to Prevent Moderate-high Recurrence and Progression Risks of Muscle-invasive Bladder Cancer
Brief Title: Transurethral Resection of Bladder Tumor (TURBT) Combined With Adjuvant Intravenous GC Chemotherapy for Non-muscle-invasive Bladder Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-SR-193
Record Dates: First submitted 2016-03-14; First posted 2016-03-23 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2015-11

CONDITIONS: Bladder Cancer; Gemcitabine and Cisplatin Chemotherapy; Epirubicin Instillation; Recurrence; Prognosis
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Monotherapy (No Intervention): Barely epirubicin was instilled after TURBT. Epirubicin was immediately instilled in 24h after TURBT. Instillation was conducted regularly for a year: once in a week for 8 times, once in two weeks for 8 times, once in a month for 6 times.
- Combination (Experimental): Patients who were pathologically confirmed as moderate-high risk NMIBC. Epirubicin was immediately instilled in 24h after TURBT and regularly conducted for a year. Intervention: GC scheme systematic chemotherapy was underwent 5 days after TURBT, which contained gemcitabine 1000-1200mg/m2. Cisplatin (70mg/m2) was intravenous dripped in the first and 8th day after TURBT. Intravenous rehydration was conducted in the second day.
  Interventions: Drug: Gemcitabine, cisplatin

INTERVENTIONS:
Drug: Gemcitabine, cisplatin — Patients who were pathologically confirmed as moderate-high risk NMIBC. Epirubicin was immediately instilled in 24h after TURBT and regularly conducted for a year. GC scheme systematic chemotherapy was underwent 5 days after TURBT, which contained gemcitabine 1000-1200mg/m2. Cisplatin (70mg/m2) was intravenous dripped in the first and 8th day after TURBT. Intravenous rehydration was conducted in the second day.
  Other Names: Combination
  Arms: Combination

SUMMARY:
It is still a challenge for urologic surgeon to prevent the post transurethral resection of bladder tumor (TURBT) recurrence of moderate-high risk non-muscle invasive bladder tumor. Adjuvant chemotherapy is a standard treatment for local progressive bladder tumor, which contains mainstream GC treatment scheme. It is common to observe clinically moderate-high risk NMIBC recurrence after routine intravesical instillation.Systematic chemotherapy can eliminate remained tumor cells especially those from mucosa basal cells so as to improve the prognosis of patients. Our clinical trial aims to investigate whether the utilization of combination of GC treatment scheme and epirubicin instillation would decrease the recurrence of moderate-high risk NMIBC.

DETAILED DESCRIPTION:
Prevention of the post-transurethral resection of bladder tumor (TURBT) recurrence of moderate-high risk non-muscle invasive bladder cancer(NMIBC) is still a difficult problem. NMIBC was classified as low, moderate and high risk patients. Moderate-high risk NMIBC contained those are multiple, recurrent, II-III grade, tumor diameter >3cm, invasive to submucosa and associated with carcinoma in situ. For those patients, no matter which treatment was conducted, for example, exchanging instillation drugs, increasing medicine dose, appending adjuvant drugs and prolonging instillation time, would not improve the prognosis of these patients. Adjuvant chemotherapy is a standard treatment for local progressive bladder tumor, which contains mainstream GC treatment scheme. For muscle invasive bladder cancer patients, radical cystectomy with neoadjuvant chemotherapy will improve patients' tumor grade and increase overall survival and disease specific survival rate.Systematic chemotherapy can eliminate remained tumor cells especially those from mucosa basal cells so as to improve the prognosis of patients. Our clinical trial aims to investigate whether the utilization of combination of GC treatment scheme and epirubicin instillation would decrease the recurrence of moderate-high risk NMIBC. In addition, we also would like to investigate the improvement of life quality after TURBT of moderate-high risk NMIBC.

ELIGIBILITY:
Inclusion Criteria:

1. moderate-high risk non-muscle invasive bladder cancer patients: Multiple,recurrent, II-III grade, tumor diameter>3cm, invasive to submucosa, associated with carcinoma in situ.
2. Normal liver and renal function.

Exclusion Criteria:

1. Liver and renal function deficiency (GFR<60ml/min*kg, ALT、AST>1.5*normal), lung function deficiency, heart failure, acute myocardial infarction, severe infection and trauma, major surgery and clinical hypotension and anaerobic conditions.
2. Attending other drug experiments.
3. Performance status, Zubrod-ECOG-WHO, ZPS≥2.
4. Pregnant.
5. Bone marrow transplantation, severe leukopenia, associated with severe infection or injury.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Tumor progression | Changes from post-chemotherapy to 5 years
Drug intervention complications | 2 years
  WBC and PLT decreasing, impaired liver function, nausea and vomiting

SECONDARY OUTCOMES:
The percent of patients transferred to radical cystectomy. | Up to 5 years
The existence of circulating tumor cells. | Before and 4 months after TURBT.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Lu, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The first affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Babjuk M, Oosterlinck W, Sylvester R, Kaasinen E, Bohle A, Palou-Redorta J, Roupret M; European Association of Urology (EAU). EAU guidelines on non-muscle-invasive urothelial carcinoma of the bladder, the 2011 update. Eur Urol. 2011 Jun;59(6):997-1008. doi: 10.1016/j.eururo.2011.03.017. Epub 2011 Mar 22. PMID 21458150
- [Result] Sylvester RJ, Oosterlinck W, Holmang S, Sydes MR, Birtle A, Gudjonsson S, De Nunzio C, Okamura K, Kaasinen E, Solsona E, Ali-El-Dein B, Tatar CA, Inman BA, N'Dow J, Oddens JR, Babjuk M. Systematic Review and Individual Patient Data Meta-analysis of Randomized Trials Comparing a Single Immediate Instillation of Chemotherapy After Transurethral Resection with Transurethral Resection Alone in Patients with Stage pTa-pT1 Urothelial Carcinoma of the Bladder: Which Patients Benefit from the Instillation? Eur Urol. 2016 Feb;69(2):231-44. doi: 10.1016/j.eururo.2015.05.050. Epub 2015 Jun 16. PMID 26091833
- [Result] Villavicencio H, Rodriguez Faba O, Palou J, Gausa L, Algaba F, Marcuello E. Bladder preservation strategy based on combined therapy in patients with muscle-invasive bladder cancer: management and results at long-term follow-up. Urol Int. 2010;85(3):281-6. doi: 10.1159/000316076. Epub 2010 Jul 30. PMID 20689253